CLINICAL TRIAL: NCT04319289
Title: Effect of Aerobic Interval Training Combined With Vitamin D Supplement on Functional Capacity and Perceived Myalgia in Middle Aged Obese Women
Brief Title: Effect of Aerobic Interval Training With Vitamin D Supplement on Functional Capacity and Perceived Myalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba Ahmed Ali Abdeen, Assistant professor, Faculty of Physical Therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020HAAE
Record Dates: First submitted 2020-03-22; First posted 2020-03-24 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group (A) (Experimental): Included 15 patients who are participating in an aerobic interval training exercise program with vitamin D supplementation (cholecalciferol 400 IU/day).
  The aerobic interval training is conducted for one hour, three days per week on a total period of 12 weeks.
  Interventions: Other: aerobic interval training and Vitamin D supplementation,
- Group (B) (Experimental): Included 15 patients who are receiving vitamin D supplementation only . One capsule containing (cholecalciferol 400 IU) was taken every day for 12 weeks
  Interventions: Drug: Vitamin D supplementation only
- Group (c) (Experimental): Included 15 patients who are participating in an aerobic interval training exercise program only. The aerobic interval training is conducted for one hour, three days per week on a total period of 12 weeks.
  Interventions: Other: aerobic interval training only

INTERVENTIONS:
Other: aerobic interval training and Vitamin D supplementation, — The participants in both groups A will be instructed to perform aerobic interval exercises at 70% maxHR for 5 minutes and then decrease activity to 50% for 5 minutes and repeat for the length of the activity (the training will be done by using bicycle ergometer(Biodex LBC, Biodex Inc., New York).• Before starting training ; Maximum heart rate calculated from the following equation: maxHR= 220-age .
  * Duration: the first five to ten minutes of each session were dedicated to warming up exercise on the bicycle in the form of slow progression exercise (to decrease the risk of hypotension, musculoskeletal injury and cardiovascular complications), followed by the active phase of exercise for 40 min., and finally cooling down phase for ten minutes. with intensity and speed decreased gradually until reaching the resting HR
  * Frequency: 3 days/week., for 12 weeks
  Also all participants in this group are taking gne capsule containing (cholecalciferol 400 IU) every day .
  Arms: Group (A)
Drug: Vitamin D supplementation only — One capsule containing (cholecalciferol 400 IU) was taken every day .
  Arms: Group (B)
Other: aerobic interval training only — The participants in group C will be instructed to perform aerobic interval exercises at 70% maxHR for 5 minutes and then decrease activity to 50% for 5 minutes and repeat for the length of the activity (the training will be done by using bicycle ergometer(Biodex LBC, Biodex Inc., New York).• Before starting training ; Maximum heart rate calculated from the following equation: maxHR= 220-age (Gellish ,2007).
  * Duration: the first five to ten minutes of each session were dedicated to warming up exercise on the bicycle in the form of slow progression exercise (to decrease the risk of hypotension, musculoskeletal injury and cardiovascular complications), followed by the active phase of exercise for 40 min., and finally cooling down phase for ten minutes. with intensity and speed decreased gradually until reaching the resting heart rate (Broderick et al.,2014).
  * Frequency: 3 days/week. The whole training lasting for 12 weeks
  Arms: Group (c)

SUMMARY:
This study aimed to investigate whether there will be an effect of adding a program of aerobic interval training in managing patients suffering from myalgia associated with vitamin D deficiency.

DETAILED DESCRIPTION:
Forty five women complaining from myalgia with vitamin D deficiency participating in this study. Their ages are ranged from 30 to 40 years.

They are assigned randomly into three groups:

* Group (A): included 15 patients who are participating in an aerobic interval training exercise program with vitamin D supplementation (cholecalciferol 400 IU/day).
* Group (B): included 15 patients who are receiving vitamin D supplementation only (cholecalciferol 400 IU/day).
* Group (C): included 15 patients who are participating in an interval training exercise program only.

The intervention will last for 12 weeks

ELIGIBILITY:
Inclusion Criteria:

* Forty five sedentry women with non specific myalgia pain.
* The patients' ages ranged from 30 -40 years.
* All patients have non specific muscle pain for more than 2 months.
* They have vitamin D deficiency.
* All patients have BMI from 25 to 34.9 kg/m2.
* All patients were clinically and medically stable when attending the study.

Exclusion Criteria:

* Unstable cardiovascular and chest problems.
* Patients with diseases which affect vitamin D level as a history of rheumatic or metabolic bone diseases and diabetes.
* Patients taking drugs which affect vitamin D level as steroids and anticonvulsants drugs .
* Musculoskeletal disorders which may affect their physical ability to do the exercises.

Ages: 30 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2020-01-12 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-05-20 (Actual)

PRIMARY OUTCOMES:
Concentration of Plasma Serum vitamin D level (25OHD) | It is performed before and after the study(12 weeks interval) for all groups
  It is performed by Laboratory BioPlex® 2200 System
Description of Functional capacity efficiency | It is performed before and after the study(12 weeks interval) for all groups
  Cooper 12-Minute Walk Test (12MWT)
Intensity of non specific muscle pain (myalgia) | It is performed before and after the study(12 weeks interval) for all groups
  A 10-cm Visual Analogue Scale (VAS) was used to evaluate the patients' pain , with 0 representing no pain and 10 representing the worst pain imaginable
Description of the improvement in Quality of life | It is performed before and after the study(12 weeks interval) for all groups
  The Short form health survey (SF-12)is often used to compare health status between groups of patients, to indentify predictors of health status

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No